CLINICAL TRIAL: NCT00069121
Title: An Open-Label Randomized Phase III Study of Intermittent Oral Capecitabine in Combination With Intravenous Oxaliplatin (Q3W) ("XELOX") Versus Fluorouracil/Leucovorin as Adjuvant Therapy for Patients Who Have Undergone Surgery for Colon Carcinoma, AJCC/UICC Stage III (Dukes Stage C)
Brief Title: A Study of Xeloda (Capecitabine) Plus Oxaliplatin in Patients With Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO16968; NCT00080691 (obsolete NCT alias)
Record Dates: First submitted 2003-09-15; First posted 2003-09-18 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Leucovorin; Fluorouracil

ARMS (2):
- 5-Fluorouracil/Leucovorin (5-FU/LV) (Active Comparator): Participants were given one of two regimens (each participating center prespecified which regimen they would use for all patients at that center): i) Mayo Clinic regimen group: LV 20 mg/m^2 IV bolus injection + 5-FU 425 mg/m^2 IV bolus injection daily on Days 1-5 of a four-week cycle, for a total of six cycles (24 weeks), or; ii) Roswell Park regimen group: LV 500 mg/m^2 by two-hour IV infusion + 5-FU 500 mg/m^2 IV bolus injection one hour after the start of the LV infusion on Day 1 of Weeks 1 to 6 of each eight-week cycle, for a total of four cycles (32 weeks).
  Interventions: Drug: Leucovorin (LV); Drug: 5-Fluorouracil (5-FU)
- Capecitabine in Combination with Oxaliplatin (XELOX) (Experimental): Capecitabine was administered as an oral twice daily outpatient intermittent treatment (3-week cycles consisting of two weeks of treatment followed by one week without treatment) combined with intravenous (IV) oxaliplatin on Day 1 of each cycle. Capecitabine was administered orally at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2) with the first dose given during the evening of Day 1 and last dose given during the morning of Day 15. Oxaliplatin was administered as a 130 mg/m^2 IV infusion over two hours on Day 1 of each cycle. The XELOX combination was administered for a total of eight cycles (24 weeks).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — 1000 milligrams per square metre of body surface area (mg/m^2) orally twice daily on days 1-15 of each 3-week cycle.
  Other Names: Xeloda
  Arms: Capecitabine in Combination with Oxaliplatin (XELOX)
Drug: Oxaliplatin — 130 mg/m^2 intravenous (IV) infusion over two hours on Day 1 of each 3-week cycle.
  Arms: Capecitabine in Combination with Oxaliplatin (XELOX)
Drug: Leucovorin (LV) — Administered by one of two regimens, as specified in the arm description.
  Arms: 5-Fluorouracil/Leucovorin (5-FU/LV)
Drug: 5-Fluorouracil (5-FU) — Administered by one of two regimens, as specified in the arm description.
  Arms: 5-Fluorouracil/Leucovorin (5-FU/LV)

SUMMARY:
This 2 arm study will compare the efficacy and safety of intermittent oral Xeloda plus Eloxatin (oxaliplatin) with that of fluorouracil/leucovorin in patients who have had surgery for colon cancer and no previous chemotherapy. Patients will be randomized to receive either 1) XELOX (Xeloda 1000mg/m2 po bid on days 1-15 + oxaliplatin) in 3 week cycles or 2)5-fluorouracil + leucovorin in 4 or 8 week cycles. The anticipated time on study treatment is until disease progression and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colon carcinoma, AJCC/UICC Stage III (Dukes stage C)
* Complete tumor resection; Patients operated with curative intent and with no macroscopic or microscopic evidence for remaining tumor who can be randomized to either treatment arm within 8 weeks after surgery. As this is an adjuvant trial patients should never have had any evidence of metastatic disease (including presence of tumor cells in the ascites).
* Have a life expectancy of at least 5 years

Exclusion Criteria:

* Pregnant or lactating women
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy, for the currently treated colon cancer
* Patients who have not completely recovered from surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1886 (Actual)
Dates: Start 2003-04-18 (Actual); Primary Completion 2011-04-21 (Actual); Study Completion 2011-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (232):
- United States (48):
  - The Cancer Center At Providence Park, Mobile, Alabama
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - Comprehensive Blood/Cancer Ctr, Bakersfield, California
  - Virginia K. Crossen Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - West Valley Hematology Oncology The Thomas and Dorothy Leavey Cancer Center, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Pomona, California
  - Sutter Cancer Center, Sacramento, California
  - Scripps Cancer Center, San Diego, California
  - Kaiser Permanente San Diego; Hepatology Research, San Diego, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - San Diego Cancer Center'S Medical Group, Vista, California
  - Innovative clinical research institute/American institute of research, Whittier, California
  - University of Colorado Health Science Center; Biomedical Research Bldg. Room 511, Aurora, Colorado
  - Hematology Oncology Associates, Fort Collins, Colorado
  - Hematology Oncology P.C., Stamford, Connecticut
  - Georgetown Uni Medical Center; Lombardi Cancer Center, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Uni of Miami School of Medicine; Sylvester Comprehensive Cancer Center, Miami, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - Hope Center, Terre Haute, Indiana
  - Ochsner Cancer Inst., New Orleans, Louisiana
  - Park Nicollet Clinic Cancer Center, Saint Louis Park, Minnesota
  - St Joseph Oncology, Saint Joseph, Missouri
  - Hematology Oncology Consultants, Inc., St Louis, Missouri
  - Hematology-Oncology Centers of the Northern Rockies, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Va Medical Center, Reno, Nevada
  - Nh Oncology Hematology, Pa, Hooksett, New Hampshire
  - Morristown Medical Center;Hematology-Oncology Assoc, Morristown, New Jersey
  - Overlook Oncology Center; Summit Medical Group, Summit, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - St. Vincent'S Hospital; Comprehensive Care Center, New York, New York
  - Presbyterian Healthcare; Cancer Research Dept, Charlotte, North Carolina
  - Moses Cone Reg Cancer Ctr, Greensboro, North Carolina
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Oncology-Hematology of Lehigh Valley, Pc, Bethlehem, Pennsylvania
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Hospital of the Uni of Pennsylvania; Section of Hematology/Oncology, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - Uni of Pittsburgh Cancer Inst. ; Oncology, Pittsburgh, Pennsylvania
  - West Clinic, Germantown, Tennessee
  - US Oncology, The Woodlands, Texas
  - Intermountain Hematology & Oncology, Salt Lake City, Utah
  - Internal Medicine Associates of Yakima Inc., Yakima, Washington
  - UNI OF WISCONSIN SCHOOL OF MEDICINE; GI Oncology Research Group, Paul P Carbone Cancer Center, Madison, Wisconsin
- Australia (7):
  - Royal Prince Alfred Hospital; Medical Oncology, Camperdown, New South Wales
  - Port Macquarie Base Hospital; Oncology, Port Macquarie, New South Wales
  - Southern Medical Day Care; Clinical Trials Unit, Wollongong, New South Wales
  - Queen Elizabeth Hospital; Medical Oncology, Woodville South, South Australia
  - Box Hill Hospital; Oncology, Box Hill, Victoria
  - Footscray Hospital, Footscray, Victoria
  - St John of God Hospital; Medical Oncology, Perth, Western Australia
- Belgium (5):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (3):
  - Hospital de Baleia; Serviço de Oncologia Clínica, Belo Horizonte, Minas Gerais
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas - FMUSP; Gastroenterologia, São Paulo, São Paulo
- Canada (23):
  - Tom Baker Cancer Centre; Dept of Medicine, Calgary, Alberta
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Bcca - Cancer Center Southern Interior, Kelowna, British Columbia
  - Bcca-Fraser Valley Cancer Centre, Surrey, British Columbia
  - Bcca - Vancouver Island Cancer Centre; Oncology, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre; Oncology, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital/Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - Hotel Dieu de Levis; Oncology, Lévis, Quebec
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Chum Campus Notre Dame, Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Hopital Du Sacre Coeur de Montreal; Pneumologie, Montreal, Quebec
  - Chuq - Hopital Hotel Dieu de Quebec; Oncology, Québec, Quebec
- China (11):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Shandong Cancer Hospital; Oncology, Shandong
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
- Finland (2):
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (4):
  - Hopital Louis Pasteur; Medecine B, Colmar
  - Hopital Claude Huriez; Medecine Interne Oncologie, Lille
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Hopital Civil; Hematologie Oncologie, Strasbourg
- Germany (4):
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Universitaetsklinikum Halle; Klinik u.Poliklinik fuer Innere Medizin IV, Halle
  - Klinikum Magdeburg gemeinnützige GmbH; Klinik Haematologie und Onkologie, Magdeburg
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
- Greece (6):
  - Evangelismos Hospital; Medical Oncology, Athens
  - Per. Gen. Hospital Ippokrateion; Oncology Dept., Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
  - Theagenio Anticancer Hospital; 3Rd Oncology Clinic, Thessaloniki
  - Theageneio Anticancer Hospital; Gastroenterology, Thessaloniki
- Queen Mary Hospital; Surgery, Hong Kong, Hong Kong
- Hungary (4):
  - Ogyi, Orszagos Gyogyszereszeti Intezet, Budapest
  - Fovarosi Szent Laszlo Korhaz-Rendelointezet; Onkologiai Osztaly X, Budapest
  - Orszagos Onkologial Intezet; Onkologiai Osztaly X, Budapest
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Ireland (3):
  - Mercy Uni Hospital; Deparment of Medical Oncology, Cork
  - St. James Hospital; Oncology, Dublin
  - Galway Uni Hospital; Oncology Dept, Galway
- Israel (12):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Rambam Medical Center; Oncology, Haifa
  - Shaare Zedek Medical Center; Oncology Dept, Jerusalem
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Nahariya Hospital; Oncology, Nahariya
  - Rabin Medical Center; Oncology Dept, Petah Tikva
  - Golda Hasharon Medical Center; Oncology, Petah Tikva
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Kaplan Medical Center; Oncology Inst., Rehovot
  - Sourasky / Ichilov Hospital; Oncology Department, Tel Aviv
  - Assaf Harofeh; Oncology, Ẕerifin
- Italy (11):
  - Ospedale Cervesi di Cattolica; ONCOLOGIA, Cattolica, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - Ospedale Degli Infermi; Divisione Di Oncologia, Rimini, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Az. Osp. Uni Ria San Martino; Cliniche Uni Rie Convenzionate U.O. Oncologia Medical, Genoa, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Ospedale Civile; Oncologia Medica, Sassari, Sardinia
  - A.O.U. Ospedali Riuniti Umberto I-G.M.Lancisi-G.Salesi Ancona;S.O.D. MED.Interna-Clinica Oncologica, Ancona, The Marches
  - Ospedale Civile; Unita Operativa Di Oncologia Medica, Livorno, Tuscany
  - Azienda Usl 7; Dept. Oncologico, Poggibonsi, Tuscany
- Mexico (4):
  - Centro Estatal de Cancerología, Chihuahua City
  - Hospital Christus Muguerza Del Parque; Centro de Rehabilitacion, Chihuahua City
  - Clinica de Especialidades # 30 Dr. Humberto Torres Sangines; Oncology, Mexicali
  - Instituto Nacional De Ciencias Medicas Y Nutricion; Nefrology, Mexico City
- New Zealand (5):
  - Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland
  - Christchurch Hospital; Dept of Oncology, Christchurch
  - Dunedin Hospital; Oncology - Haematology Clinical Practice Group, Dunedin
  - Palmerston North Hospital; Regional Cancer Treatment Service, Palmerston North
  - Wellington Hospital; Regional Oncology Unit, Wellington
- Isthmian Medical Research Center, S.A.; Oncology, Panama City, Panama
- Poland (6):
  - Rydygiera Hospital; Chemotherapy, Krakow
  - Wojewodzki Szpital Specjalistyczny Im. M. Kopernika; Oddzial Chorob Rozrostowych, Lodz
  - Wielkopolskie Centrum Onkologii; Oddzial Chemioterapii, Poznan
  - Zachodniopomorskie Centrum Onkologii, Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Klinika Nowotworow Jelita Grubego, Warsaw
  - Lubuski Osrodek Onkologii, Szpital Wojewodzki; Oddzial Onkologii, Zielona Góra
- Portugal (3):
  - Hospital Jose Joaquim Fernandes; Unidade de Oncologia Medica, Beja
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Russia (4):
  - N.N.Burdenko Main Military Clinical Hospital; Chemotherapy, Moscow
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - Petrov Research Inst. of Oncology; Dept of Bio-Therapy & Transplantation of Bone Marrow, Saint Petersburg
  - St. Petersburg City Clinical Oncological Dispensary; Colorectal (Department 4), Saint Petersburg
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- South Africa (5):
  - Panorama Medical Clinic; Oncology Unit, Cape Town
  - Hopelands Cancer Centre; Oncology, Durban
  - Hopelands Cancer Centre ST. ANNES HOSPITAL; DEPT. OF ONCOLOGY, Pietermaritzburg
  - Little Company of Mary Hospital; Mary Potter Oncology Centre, Pretoria
  - Sandton Oncology Medical Group, Sandton
- South Korea (5):
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei Medical Center; Dept. of Medicine , Division of Hemato-Oncology, Seoul
  - Hanyang Uni Hospital; Dept. of Internal Medicine , Section of Hemato-Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
- Spain (20):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital Severo Ochoa; Servicio de Oncologia, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitario de la Princesa; Servicio de Oncologia, Madrid
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
- Universitaetsspital Basel; Onkologie, Basel, Switzerland
- Taiwan (3):
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Mackay Memorial Hospital; Department of Surgery, Division of Colon and Rectal Surgery, Taipei
  - Chang Gung Medical Foundation - Linkou; Colo-rectal Surgery, Taoyuan District
- Thailand (5):
  - Bumrungrad Hospital Foundation; Horizon Centre, Bangkok
  - Pramongkutklao Hospital; Medicine - Medical Oncology Unit, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Srinagarind Hospital; Medical Oncology Unit, Khon Kaen
- United Kingdom (24):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - The Royal Sussex County Hospital; the Sussex Cancer Centre, Brighton
  - West Suffolk Hospital Nhs Trust; Gi Corridor, Bury St Edmunds
  - Addenbrooke'S Hospital; Univ.Dept.& Mrc Unit of Clin.Oncology & Radiotherapeutics, Cambridge
  - Derbyshire Royal Infirmary; Dept of Oncology, Derby
  - Cruk Clinical Trials Unit; Level 0 Beatson West Of Scotland Cancer Ctr, Glasgow
  - Royal Surrey County Hospital; St. Lukes Cancer Centre, Guildford
  - St James Institute of Oncology, Leeds
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - St Thomas Hospital; Oncology Dept, London
  - Royal Marsden Nhs Trust; Consultant Cancer Physician, London
  - Hammersmith Hospital; Mrc Clinical Science Centre, London
  - Charing Cross Hospital; Medical Oncology., London
  - Maidstone Hospital, Maidstone
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - James Cook Uni Hospital, Middlesbrough
  - Northern Centre for Cancer Care;Oncology, Newcastle upon Tyne
  - Mount Vernon Hospital; Centre For Cancer Treatment, Northwood
  - Nottingham City Hospital; Oncology, Nottingham
  - Derriford Hospital; Plymouth Oncology Centre, Plymouth
  - North Wales Cancer Treatment Centre, Glan Clwyd Hospital, Rhyl
  - Salisbury District General Hospital; Medical Oncology Dept, Salisbury
  - Southampton General Hospital; Somers Cancer Research Building, Southampton
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Schmoll HJ, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Hoersch S, Rittweger K, Haller DG. Capecitabine Plus Oxaliplatin Compared With Fluorouracil/Folinic Acid As Adjuvant Therapy for Stage III Colon Cancer: Final Results of the NO16968 Randomized Controlled Phase III Trial. J Clin Oncol. 2015 Nov 10;33(32):3733-40. doi: 10.1200/JCO.2015.60.9107. Epub 2015 Aug 31. PMID 26324362

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-FU/LV: Given by one of two regimens. • Mayo Clinic regimen group: LV 20 mg/m^2 IV bolus injection + 5-FU 425 mg/m^2 IV bolus injection daily on Days 1-5 of a four-week cycle, for a total of six cycles (24 weeks), or • Roswell Park regimen group: LV 500 mg/m^2 by two-hour IV infusion + 5-FU 500 mg/m^2 IV bolus injection one hour after the start of the LV infusion on Day 1 of Weeks 1 to 6 of each eight-week cycle, for a total of four cycles (32 weeks)
- XELOX: Capecitabine administered as an oral twice daily outpatient intermittent treatment (3-week cycles consisting of two weeks of treatment followed by one week without treatment) combined with intravenous (IV) oxaliplatin on Day 1 of each cycle. Capecitabine was administered orally at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2) with the first dose given during the evening of Day 1 and last dose given during the morning of Day 15. Oxaliplatin was administered as a 130 mg/m^2 IV infusion over two hours on Day 1 of each cycle. The XELOX combination was administered for a total of eight cycles (24 weeks)
Period: Overall Study
Arm/Group | 5-FU/LV | XELOX
Started | 942 | 944
Received Treatment | 926 (Safety Population) | 938 (Safety Population)
Completed | 575 (total includes Completed and Alive in follow-up) | 619 (total includes Completed and Alive in follow-up)
Not Completed | 367 | 325
Not completed — Death | 286 | 242
Not completed — Withdrawal by Subject | 18 | 20
Not completed — Lost to Follow-up | 63 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-FU/LV | XELOX | Total
Number analyzed (Participants) | 942 | 944 | 1886
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.76) | 59.8 (10.95) | 60.2 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 442 | 431 | 873
  Male | 500 | 513 | 1013
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 442 | 431 | 873
  Male | 500 | 513 | 1013

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) [Number of Events]
Description: Determination of an event was based on tumor assessments and survival follow-up assessments. A disease-free survival (DFS) event was defined as any recurrence of the original colon cancer or appearance of a new colon or rectal cancer (proven by cytology or histology, when possible) or death due to any cause, whichever was earliest. Participants who had not had any such event at the time of data analysis were censored at the last date they were known to be event-free. Participants with no tumor assessments after baseline were censored at Day 1. An isolated event of increased CEA, or unexplained clinical deterioration were not considered to be evidence of relapse without support of other objective measurements. The date of relapse was defined as the date of the definitive assessment by objective measurements.
Time Frame: Time from randomization date to date of first DFS event/date last known to be event-free. Median observation time for DFS was 74 months (range: 0-95 months).
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
Participants
  Patients with Event | 379 | 320
  Patients without Events | 563 | 624

2. Secondary Outcome: Relapse-Free Survival (RFS) [Number of Events]
Description: A relapse-free survival (RFS) event included recurrence of the original colon cancer, development of a new colon or rectal cancer, and deaths related to any of the following: treatment, recurrence of the original colon cancer, or development of a new colon or rectal cancer. Participants who had not had any such event at the time of data analysis were censored at the last date they were known to be event-free. Participants whose cause of death was unrelated to treatment or disease recurrence were censored at the time of the last tumor assessment.
Time Frame: Time from randomization date to date of first RFS event/date last known to be event-free. Median observation time for RFS was 74 months (range: 0-95 months).
Population: Intent-to-Treat (ITT) Population: all randomized participants who gave written informed consent. Participants in the ITT population were analyzed according to the treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
Participants
  Patients With Event | 356 | 290
  Patients Without Events | 586 | 654

3. Primary Outcome: Disease-Free Survival (DFS) [Time to Event]
Description: Determination of an event was based on tumor assessments and survival follow-up assessments. A disease-free survival (DFS) event was defined as any recurrence of the original colon cancer or appearance of a new colon or rectal cancer (proven by cytology or histology, when possible) or death due to any cause, whichever was earliest. Participants who had not had any such event at the time of data analysis were censored at the last date they were known to be event-free. Participants with no tumor assessments after baseline were censored at Day 1. An isolated event of increased CEA, or unexplained clinical deterioration were not considered to be evidence of relapse without support of other objective measurements. The date of relapse was defined as the date of the definitive assessment by objective measurements. The median was estimated by the Kaplan-Meier method. The full range values include censored observations.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
months | NA [0 to 95] — The median time for DFS was not reached in this adjuvant trial; however, due to a late event in the XELOX arm and an artificial drop in the Kaplan-Meier estimate, an artificial median estimate for the XELOX groups appears. | 88.6 [0 to 89]
Statistical Analysis 1: Comparison: 5-FU/LV vs XELOX; Test type: Superiority; p = 0.0038, Log Rank — This test used a two-sided significance level of 5%; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.69 to 0.93] — The hazard ratio was calculated as XELOX versus 5-FU/LV arms

4. Secondary Outcome: Relapse-Free Survival (RFS) [Time to Event]
Description: A relapse-free survival (RFS) event included recurrence of the original colon cancer, development of a new colon or rectal cancer, and deaths related to any of the following: treatment, recurrence of the original colon cancer, or development of a new colon or rectal cancer. Participants who had not had any such event at the time of data analysis were censored at the last date they were known to be event-free. Participants whose cause of death was unrelated to treatment or disease recurrence were censored at the time of the last tumor assessment. The median was estimated by the Kaplan-Meier method. The full range values include censored observations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
months | NA [0 to 95] — The median time for RFS was not reached in this adjuvant trial; however, due to a late event in the XELOX arm and an artificial drop in the Kaplan-Meier estimate, an artificial median estimate for the XELOX groups appears. | 88.6 [0 to 89]
Statistical Analysis 1: Comparison: 5-FU/LV vs XELOX; Test type: Other — Descriptive analysis only; p = 0.0015, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.67 to 0.91] — The hazard ratio was calculated as XELOX versus 5-FU/LV arms

5. Secondary Outcome: Overall Survival [Number of Events]
Description: Overall survival was measured as the time from randomization to the date of death, irrespective of the cause of death. Participants who were not reported as having died at the time of the analysis were censored using the date they were last known to be alive.
Time Frame: Time from randomization date to date of death/date last known to be alive. Median observation time was 83 months (range: 0-95 months).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
Participants
  Patients With Event | 286 | 242
  Patients Without Events | 656 | 702

6. Secondary Outcome: Overall Survival [Time to Event]
Description: Overall survival was measured as the time from randomization to the date of death, irrespective of the cause of death. Participants who were not reported as having died at the time of the analysis were censored using the date they were last known to be alive. The median was estimated by the Kaplan-Meier method. The full range values include censored observations.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | 5-FU/LV | XELOX
Number analyzed (Participants) | 942 | 944
months | NA [0 to 95] — The median time to death was not reached in this adjuvant trial. | NA [0 to 93] — The median time to death was not reached in this adjuvant trial.
Statistical Analysis 1: Comparison: 5-FU/LV vs XELOX; Test type: Other — Descriptive analysis only; p = 0.0367, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.99] — The hazard ratio was calculated as XELOX versus 5-FU/LV arms

7. Secondary Outcome: Number of Participants With at Least One Adverse Event by Most Severe Intensity
Description: The intensity of all adverse events (AEs) was categorized according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) (version 3.0) grading system. If an AE had occurred which was not contained in the NCI-CTC, a four-point scale (mild, moderate, severe, life-threatening) was used. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Only the most severe intensity was counted for multiple occurrences of an AE in one individual. See the AEs results table for details.
Time Frame: From time of very first drug intake to 28 days after very last drug intake (median [full range] duration of study treatment per arm: 5-FU/LV MAYO CLINIC: 145 [4-208] days; 5-FU/LV ROSWELL PARK: 204 [1-239] days; XELOX: 163 [1-275] days).
Population: Safety Population: all participants who were randomized and did receive at least one dose of capecitabine, 5-FU, or oxaliplatin. Participants in the safety population were analyzed according to the study treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- 5-FU/LV MAYO CLINIC: Mayo Clinic regimen group: LV 20 mg/m^2 IV bolus injection + 5-FU 425 mg/m^2 IV bolus injection daily on Days 1-5 of a four-week cycle, for a total of six cycles (24 weeks)
- 5-FU/LV ROSWELL PARK: Roswell Park regimen group: LV 500 mg/m^2 by two-hour IV infusion + 5-FU 500 mg/m^2 IV bolus injection one hour after the start of the LV infusion on Day 1 of Weeks 1 to 6 of each eight-week cycle, for a total of four cycles (32 weeks)
Arm/Group | 5-FU/LV MAYO CLINIC | 5-FU/LV ROSWELL PARK | XELOX
Number analyzed (Participants) | 657 | 269 | 938
Participants
  Mild AEs | 557 | 256 | 855
  Moderate AEs | 493 | 217 | 792
  Severe AEs | 299 | 146 | 548
  Life-Threatening | 83 | 21 | 63

ADVERSE EVENTS:
Time Frame: From time of very first drug intake to 28 days after very last drug intake (median [full range] duration of study treatment per arm: 5-FU/LV MAYO CLINIC: 145 [4-208] days; 5-FU/LV ROSWELL PARK: 204 [1-239] days; XELOX: 163 [1-275] days).
Description: AE reporting is based on the Safety Analysis Population; the patients who were randomized and received at least one dose of capecitabine, 5-FU, or oxaliplatin. Safety Population 5-FU/LV (n = 926); XELOX (n = 938)
Groups:
- 5-FU/LV MAYO CLINIC; 5-FU/LV ROSWELL PARK: 5-fluorouracil/leucovorin
- XELOX: Capecitabine in Combination with Intravenous Oxaliplatin (Q3W)
Arm/Group | 5-FU/LV MAYO CLINIC | 5-FU/LV ROSWELL PARK | XELOX
All-Cause Mortality (participants affected / at risk) | 215/664 | 71/278 | 242/944
Serious Adverse Events (participants affected / at risk) | 134/657 | 88/269 | 208/938
Other Adverse Events (participants affected / at risk) | 622/657 | 262/269 | 926/938
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU/LV MAYO CLINIC (N=657) | 5-FU/LV ROSWELL PARK (N=269) | XELOX (N=938)
DIARRHOEA (Gastrointestinal disorders) | 39 | 24 | 55
STOMATITIS ALL (Gastrointestinal disorders) | 22 | 0 | 2
VOMITING (Gastrointestinal disorders) | 6 | 3 | 15
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 3 | 13
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 5 | 2 | 7
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 3 | 8
ILEUS (Gastrointestinal disorders) | 2 | 4 | 3
NAUSEA (Gastrointestinal disorders) | 3 | 1 | 4
COLITIS (Gastrointestinal disorders) | 1 | 1 | 3
ENTERITIS (Gastrointestinal disorders) | 2 | 2 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 4
SUBILEUS (Gastrointestinal disorders) | 1 | 0 | 3
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 | 1 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 1
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 0 | 0 | 2
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 2
ILEITIS (Gastrointestinal disorders) | 0 | 0 | 2
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 0 | 2
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1 | 0
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 | 1 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0
CAECITIS (Gastrointestinal disorders) | 0 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 1
COLONIC FISTULA (Gastrointestinal disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL OEDEMA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1 | 0
INTERNAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
MECHANICAL ILEUS (Gastrointestinal disorders) | 0 | 0 | 1
OESOPHAGEAL MASS (Gastrointestinal disorders) | 0 | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 1 | 0 | 0
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 0 | 0 | 1
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 1 | 5
SEPSIS (Infections and infestations) | 3 | 1 | 3
NEUTROPENIC SEPSIS (Infections and infestations) | 5 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 2 | 1
BACTERAEMIA (Infections and infestations) | 0 | 0 | 3
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 1 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 2
INFECTION (Infections and infestations) | 0 | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
ENDOPHTHALMITIS (Infections and infestations) | 0 | 1 | 0
HEPATITIS B (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
SEPSIS SYNDROME (Infections and infestations) | 0 | 1 | 0
SKIN INFECTION (Infections and infestations) | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 31 | 2 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 8 | 2 | 3
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 10 | 24
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 3 | 5
HYPOTENSION (Vascular disorders) | 0 | 1 | 2
THROMBOSIS (Vascular disorders) | 1 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 2
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0 | 1
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 0 | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0
NECROSIS OF ARTERY (Vascular disorders) | 1 | 0 | 0
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 2 | 3 | 12
CHEST PAIN (General disorders) | 0 | 1 | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 2
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
DYSAESTHESIA PHARYNX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1 | 5
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 3
ANGINA PECTORIS (Cardiac disorders) | 2 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 1
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 2 | 1 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 3
DIZZINESS (Nervous system disorders) | 1 | 0 | 1
CEREBRAL AMYLOID ANGIOPATHY (Nervous system disorders) | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 1
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1
HEMIPLEGIA (Nervous system disorders) | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 1 | 0 | 0
SUPERIOR SAGITTAL SINUS THROMBOSIS (Nervous system disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 0 | 3
HAEMATURIA (Renal and urinary disorders) | 1 | 1 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1
UROGENITAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 0 | 1
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 3 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
HEPATIC LESION (Hepatobiliary disorders) | 0 | 0 | 1
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 2
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1
ANAPHYLACTOID REACTION (Immune system disorders) | 0 | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
INTERVERTEBRAL DISC DISPLACEMENT (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 0 | 1 | 0
BLOOD BILIRUBIN ABNORMAL (Investigations) | 0 | 0 | 1
CULTURE STOOL POSITIVE (Investigations) | 0 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1
OVARIAN MASS (Reproductive system and breast disorders) | 1 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0 | 0
EYE MOVEMENT DISORDER (Eye disorders) | 0 | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU/LV MAYO CLINIC (N=657) | 5-FU/LV ROSWELL PARK (N=269) | XELOX (N=938)
DIARRHOEA (Gastrointestinal disorders) | 449 | 219 | 577
NAUSEA (Gastrointestinal disorders) | 350 | 190 | 625
STOMATITIS ALL (Gastrointestinal disorders) | 419 | 57 | 195
VOMITING (Gastrointestinal disorders) | 142 | 103 | 415
ABDOMINAL PAIN (Gastrointestinal disorders) | 118 | 92 | 204
CONSTIPATION (Gastrointestinal disorders) | 82 | 48 | 187
DYSPEPSIA (Gastrointestinal disorders) | 38 | 37 | 87
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 44 | 21 | 77
FLATULENCE (Gastrointestinal disorders) | 21 | 29 | 47
DRY MOUTH (Gastrointestinal disorders) | 23 | 14 | 26
PARAESTHESIA (Nervous system disorders) | 16 | 10 | 339
NEUROPATHY PERIPHERAL (Nervous system disorders) | 8 | 12 | 279
DYSGEUSIA (Nervous system disorders) | 86 | 40 | 126
HEADACHE (Nervous system disorders) | 46 | 31 | 103
DIZZINESS (Nervous system disorders) | 34 | 34 | 99
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 | 11 | 152
DYSAESTHESIA (Nervous system disorders) | 1 | 1 | 104
LETHARGY (Nervous system disorders) | 46 | 3 | 52
HYPOAESTHESIA (Nervous system disorders) | 2 | 7 | 59
FATIGUE (General disorders) | 148 | 170 | 332
ASTHENIA (General disorders) | 91 | 44 | 167
PYREXIA (General disorders) | 60 | 43 | 108
TEMPERATURE INTOLERANCE (General disorders) | 0 | 1 | 104
OEDEMA PERIPHERAL (General disorders) | 22 | 29 | 51
CHILLS (General disorders) | 9 | 16 | 29
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 56 | 42 | 278
ALOPECIA (Skin and subcutaneous tissue disorders) | 159 | 25 | 40
RASH (Skin and subcutaneous tissue disorders) | 65 | 41 | 84
DRY SKIN (Skin and subcutaneous tissue disorders) | 41 | 44 | 45
PRURITUS (Skin and subcutaneous tissue disorders) | 20 | 17 | 21
NEUTROPENIA (Blood and lymphatic system disorders) | 232 | 36 | 260
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 4 | 167
ANAEMIA (Blood and lymphatic system disorders) | 32 | 36 | 64
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 36 | 3 | 4
ANOREXIA (Metabolism and nutrition disorders) | 101 | 77 | 240
DEHYDRATION (Metabolism and nutrition disorders) | 24 | 33 | 68
HYPOKALAEMIA (Metabolism and nutrition disorders) | 20 | 33 | 58
DECREASED APPETITE (Metabolism and nutrition disorders) | 16 | 15 | 27
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 | 35 | 47
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 39 | 20 | 38
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 | 16 | 63
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 24 | 30 | 40
DYSAESTHESIA PHARYNX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 93
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 20 | 24
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 17 | 21 | 117
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22 | 26 | 41
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 | 25 | 46
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 55
INSOMNIA (Psychiatric disorders) | 49 | 38 | 78
ANXIETY (Psychiatric disorders) | 22 | 31 | 49
DEPRESSION (Psychiatric disorders) | 14 | 24 | 35
NASOPHARYNGITIS (Infections and infestations) | 20 | 15 | 32
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 18 | 29
URINARY TRACT INFECTION (Infections and infestations) | 14 | 20 | 22
LACRIMATION INCREASED (Eye disorders) | 53 | 49 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.